CLINICAL TRIAL: NCT01722305
Title: Phase I Trial of Pomalidomide for Patients With Relapsed/Refractory Primary CNS Lymphoma and Primary Vitreoretinal Lymphoma
Brief Title: Pomalidomide and Dexamethasone in Treating Patients With Relapsed or Refractory Primary Central Nervous System Lymphoma or Newly Diagnosed or Relapsed or Refractory Intraocular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1281; NCI-2012-01948 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1281 (Other: Mayo Clinic in Florida); P30CA015083 (NIH)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Burkitt Lymphoma; Central Nervous System Lymphoma; Intraocular Lymphoma; Primary Diffuse Large B-Cell Lymphoma of the Central Nervous System; Recurrent Adult Diffuse Large Cell Lymphoma; Retinal Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Intraocular Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pomalidomide, dexamethasone) (Experimental): Patients receive pomalidomide PO on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22 of courses 1 and 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacological Study — Optional correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase I trial studies the side effects and best dose of pomalidomide when given together with dexamethasone in treating patients with primary central nervous system lymphoma that has come back (relapsed) or does not respond to treatment (refractory) or intraocular lymphoma that is newly diagnosed, relapsed or refractory. Pomalidomide may stimulate the immune system to kill cancer cells. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, stopping them from dividing, or by stopping them from spreading. Giving pomalidomide together with dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of pomalidomide in combination with dexamethasone in patients with relapsed/refractory primary central nervous system lymphoma (PCNSL) or primary vitreoretinal lymphoma (PVRL).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy (overall response rate) and safety of pomalidomide in combination with dexamethasone in patients with PCNSL and PVRL lymphoma in an MTD expanded cohort.

II. To evaluate overall survival and progression free survival.

TERTIARY OBJECTIVES:

I. To study the pharmacokinetics of pomalidomide in the central nervous system. II. To identify the predictive biomarkers for responsiveness to pomalidomide.

OUTLINE: This is a dose-escalation study of pomalidomide.

Patients receive pomalidomide orally (PO) on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22 of courses 1 and 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory primary central nervous system (CNS) diffuse large B cell lymphoma (PCNSDLBCL) with a CNS lesion, with cerebrospinal fluid (CSF) relapse with positive CSF cytology, or with ocular relapse with positive ocular tissue biopsy; NOTE: tissue biopsy is not absolutely necessary for CNS tumor unless clinical and radiologic findings strongly suggest other etiologies as per treating physician; initial diagnosis must be made by tissue biopsy; NOTE: patients with B-cell lymphoma with features intermediate between diffuse large B-cell lymphoma and Burkitt lymphoma are also eligible for the protocol as long as they meet other criteria; patients with typical Burkitt lymphoma are not eligible
* Relapsed/refractory primary vitreoretinal diffuse large B cell lymphoma (DLBCL) with a CNS lesion, with CSF relapse with positive CSF cytology, or with ocular relapse with positive ocular tissue biopsy; NOTE: tissue biopsy requirement of the CNS lesion is as outlined in bullet above
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2 or 3
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets (PLT) >= 100,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN the direct bilirubin must be =< 1.5 x ULN (=< 0.45 mg/dL)
* Aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine =< 2.5 x ULN
* Females of reproductive potential must be willing to adhere to the scheduled pregnancy testing as required in the POMALYST REMS (TM) program
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or heparin)
* Provide informed written consent
* Willing to return to participating medical institutions for follow-up
* Willing to provide tissue samples for correlative research purposes
* Willing to be registered into the mandatory POMALYST REMS (TM) program, and willing and able to comply with the requirements of the POMALYST REMS (TM) program

Exclusion Criteria:

* Any of the following

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Uncontrolled infection
* Therapy with myelosuppressive chemotherapy or biologic therapy < 21 days prior to registration; NOTE: patients who have recovered from cytopenia related to previous treatment and meet criteria of this protocol will be eligible
* Persistent toxicities >= grade 3 from prior chemotherapy or biological therapy regardless of interval since last treatment
* History of thromboembolic episodes =< 3 months prior to registration
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Immunodeficiency states including human immunodeficiency virus (HIV) infection
* Active hepatitis B or C with uncontrolled disease; NOTE: a detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients; hepatitis B core immunoglobulin M antibody (HBcIgM Ab), hepatitis B surface antigen (HBsAg) and hepatitis C antibody screen (HCV Ab Scrn) w/reflex testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior hepatitis B (HBV) infection
* Active other malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment
* Inability to swallow or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) that would preclude use of oral medications
* Any severe and/or uncontrolled medical conditions or other conditions that, in the treating physician's opinion, could adversely impact their ability to participate in the study
* Major surgery =< 4 weeks prior to registration or have not recovered from side effects of such therapy
* New York Heart Association classification III or IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
MTD of pomalidomide when given in combination with dexamethasone determined by dose-limiting toxicities graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | 28 days
  The number and severity of all adverse events will be tabulated and summarized in this patient population both overall and by dose level. The grade 3+ adverse events will also be described and summarized in a similar fashion. Overall toxicity incidence as well as toxicity profiles by dose level and patient will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.

SECONDARY OUTCOMES:
Incidence of adverse events, graded according to CTCAE 4.0 | Up to 30 days post-treatment
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.
Overall response rate defined as number of patients with an objective status of complete response (CR), complete response/unconfirmed (Cru), or partial response (PR) divided by total number of evaluable patients | Up to 2 years
  Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Overall survival time | Time from registration to death due to any cause, assessed up to 2 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Progression-free survival | Time from registration to progression or death due to PCNSL or PVRL lymphoma, assessed up to 2 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.

OTHER OUTCOMES:
Pharmacokinetics of pomalidomide in the CNS | Up to day 22 of course 1
  Based on pomalidomide levels in blood and CSF at different time points, area under curve will be determined.
Predictive biomarkers for response to pomalidomide | Up to day 21 of course 1
  Correlation studies will be performed to identify predictive immune markers for response to pomalidomide. Immune cell counts and cytokine profile will be evaluated in blood and CSF at day 1 and day 21 of course 1. Values at each time point and changes after pomalidomide treatment will be both graphically and quantitatively summarized and explored. Wilcoxon rank sum test and Fisher's exact test will be utilized where appropriate to assess the relationships of these markers with response.

CONTACTS AND LOCATIONS:
Overall Officials: Han Tun, Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Tun HW, Johnston PB, DeAngelis LM, Atherton PJ, Pederson LD, Koenig PA, Reeder CB, Omuro AMP, Schiff D, O'Neill B, Pulido J, Jaeckle KA, Grommes C, Witzig TE. Phase 1 study of pomalidomide and dexamethasone for relapsed/refractory primary CNS or vitreoretinal lymphoma. Blood. 2018 Nov 22;132(21):2240-2248. doi: 10.1182/blood-2018-02-835496. Epub 2018 Sep 27. PMID 30262659